CLINICAL TRIAL: NCT07370740
Title: A Randomized, Double-blind, Placebo-controlled, Parallel Clinical Trial to Investigate the Safety and Efficacy of Bloat on Gas and Bloating in Healthy Women
Brief Title: A Clinical Trial to Investigate the Safety and Efficacy of Bloat on Gas and Bloating in Healthy Women
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Arrae (Industry)
Collaborators: KGK Science Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 25ARCCB01
Record Dates: First submitted 2026-01-12; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Bloating; Gastrointestinal Symptoms; Intestinal Gas
Keywords: Bloat; Arrae; Bloating; Intestinal Gas; Gastrointestinal symptoms
MeSH Terms: interventions — Poloxalene

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bloat (Experimental): Bloat is comprised of a novel combination of ginger root extract, bromelain, peppermint leaf extract, dandelion root extract, lemon balm herb top extract, and slippery elm inner bark extract.
  Interventions: Dietary Supplement: Bloat
- Placebo (Placebo Comparator): Placebo is comprised of white rice flour
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Bloat — Participants will be instructed to take one dose (2 capsules) 30 minutes after consumption of the entire standardized meal during the screening/baseline clinic visit.
  Arms: Bloat
Other: Placebo — Participants will be instructed to take one dose (2 capsules) 30 minutes after consumption of the entire standardized meal during the screening/baseline clinic visit
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to investigate the safety and efficacy of Bloat on gas and bloating in healthy women. The main question it aims to answer is what is the change in postprandial gas and bloating from pre-dose at t = 60 mins post-dose between Bloat and placebo, as assessed by Gas and Bloating Likert scale at screening/baseline.

Participants will be asked to consume one dose of Bloat or Placebo and answer questionnaires on gas and bloating.

ELIGIBILITY:
Inclusion Criteria:

1. Females aged 18-65 years, inclusive
2. Females not of child-bearing potential, defined as those who have undergone a sterilization procedure (e.g. hysterectomy, bilateral oophorectomy, bilateral tubal ligation, complete endometrial ablation) or have been post-menopausal for at least one year prior to screening Or,

   Individuals of child-bearing potential must have a negative baseline urine pregnancy test and agree to use a medically approved method of birth control for the duration of the study. All hormonal birth control must have been in use for a minimum of 3 months. Acceptable methods of birth control include:
   * Hormonal contraceptives including oral contraceptives, hormone birth control patch (Ortho Evra), vaginal contraceptive ring (NuvaRing), injectable contraceptives (Depo-Provera, Lunelle), or hormone implant (Norplant System)
   * Double-barrier method
   * Intrauterine devices
   * Non-heterosexual lifestyle and agrees to use contraception if planning on changing to heterosexual partner(s)
   * Vasectomy of partner at least 6 months prior to screening
   * Abstinence and agrees to use contraception if planning on becoming sexually active during the study
3. Recurrent bloating and/or distension occurring on average at least one day per week which predominates over other GI symptoms as assessed by the QI
4. Experiences significant gas and bloating after consumption of the standardized meal provided at screening/baseline, as assessed by a score of 0 (absent) or 1 (mild) pre-meal and a score of 2 (moderate) or 3 (severe) post-meal
5. Agrees to maintain current lifestyle habits (diet, physical activity, medications, supplements, and sleep) as much as possible throughout the study
6. Provided voluntary, written, informed consent to participate in the study
7. Healthy as determined by medical history as assessed by Qualified Investigator

Exclusion Criteria:

1. Individuals who are pregnant, breast feeding, or planning to become pregnant during the study
2. Participants residing in the same household as another study participant unless they are enrolled consecutively (e.g. not actively enrolled at the same time)
3. Allergy, sensitivity, intolerance, or dietary restriction preventing consumption of IP, placebo, or standardized meal ingredients
4. Current or history of any significant diseases of the GI tract or digestive disorders (e.g., irritable bowel syndrome, celiac disease, inflammatory bowel disease, functional constipation, gastroesophageal reflux disease, being treated within the past year for H. pylori infection or gastric ulcer) as assessed by the QI
5. Unstable metabolic disease or chronic diseases as assessed by the QI
6. Unstable hypertension. Treatment on a stable dose of medication for at least 3 months will be considered by the QI
7. Type I or Type II diabetes
8. Significant cardiovascular event in the past 6 months. Participants with no significant cardiovascular event on stable medication may be included after assessment by the QI on a case-by-case basis
9. History of or current diagnosis with kidney and/or liver diseases as assessed by the QI on a case-by-case basis, with the exception of history of kidney stones in participants who are symptom free for 6 months
10. Self-reported confirmation of current or pre-existing thyroid condition. Treatment on a stable dose of medication for at least 3 months will be considered by the QI
11. Major surgery in the past 3 months or individuals who have planned surgery during the course of the study. Participants with minor surgery will be considered on a case-by-case basis by the QI
12. Cancer, except skin basal cell carcinoma completely excised with no chemotherapy or radiation with a follow up that is negative. Volunteers with cancer in full remission for more than five years after diagnosis are acceptable
13. Individuals with an autoimmune disease or are immune compromised as assessed by the QI
14. Chronic use of cannabinoid products (>2 times/week) as assessed by the QI. Occasional users will be required to washout and abstain for the duration of the study period
15. Regular use of tobacco or nicotine products in the past 6 months, as assessed by the QI. Occasional users will be required to washout and abstain for the duration of the study period
16. Alcohol intake average of >2 standard drinks per day as assessed by the QI
17. Alcohol or drug abuse within the last 12 months
18. Current use of prescribed and/or over-the-counter (OTC) medications, supplements, and/or consumption of food/drinks that may impact the efficacy and/or safety of the IP (Section 7.3)
19. Participation in other clinical research studies 30 days prior to baseline, as assessed by the QI
20. Individuals who are unable to give informed consent
21. Any other condition or lifestyle factor, that, in the opinion of the QI, may adversely affect the participant's ability to complete the study or its measures or pose significant risk to the participant

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 100 (Estimated)
Dates: Start 2026-05 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
The difference in change in postprandial gas and bloating from pre-dose at t = 60 mins post-dose between Bloat and placebo | Day 0 to 56
  The difference in change in postprandial gas and bloating from pre-dose at t = 60 mins post-dose between Bloat and placebo, as assessed by Gas and Bloating Likert scale at screening/baseline. On a scale of 0 to 3, with 0 being "mild" and 3 being "severe".

SECONDARY OUTCOMES:
The difference in change in GI symptoms from baseline between Bloat and placebo | Day 0 to 28
  The difference in change in GI symptoms from baseline at Day 28 between Bloat and placebo, as assessed by PROMIS-GI Gas and Bloating Scale. On a scale of 0 to 4, with 0 being "no symptoms" to 4 being "severe symptoms"
The difference in change in GI symptoms from baseline between Bloat and placebo | Day 0 to 56
  The difference in change in GI symptoms from baseline at Day 56 between Bloat and placebo, as assessed by PROMIS-GI Gas and Bloating Scale. On a scale of 0 to 4, with 0 being "no symptoms" to 4 being "severe symptoms"
The difference in change in GI symptoms from baseline between Bloat and placebo | Day 0 to 28
  The difference in change in GI symptoms from baseline at Day 28 between Bloat and placebo, as assessed by PROMIS-GI Reflux Scale. On a scale of 0 to 4, with 0 being "no symptoms" to 4 being "severe symptoms"
The difference in change in GI symptoms from baseline between Bloat and placebo | Day 0 to 56
  The difference in change in GI symptoms from baseline at Day 56 between Bloat and placebo, as assessed by PROMIS-GI Reflux Scale. On a scale of 0 to 4, with 0 being "no symptoms" to 4 being "severe symptoms"
The difference in change in GI symptoms from baseline between Bloat and placebo | Day 0 to 28
  The difference in change in GI symptoms from baseline at Day 28 between Bloat and placebo, as assessed by PROMIS- GI Belly Pain Scale. On a scale of 0 to 4, with 0 being "no symptoms" to 4 being "severe symptoms"
The difference in change in GI symptoms from baseline between Bloat and placebo | Day 0 to 56
  The difference in change in GI symptoms from baseline at Day 56 between Bloat and placebo, as assessed by PROMIS- GI Belly Pain Scale. On a scale of 0 to 4, with 0 being "no symptoms" to 4 being "severe symptoms"
The difference in change in gas and bloating scores as assessed weekly by the Gas and Bloating Likert scales | Day 0 to 56
  The difference in change in gas and bloating scores as assessed weekly by the Gas and Bloating Likert scales. On a scale of 0 to 4, with 0 being "no symptoms" to 4 being "severe symptoms".

CONTACTS AND LOCATIONS:
Overall Officials: David Crowley, MD, Principal Investigator — KGK Science Inc.
Locations (1):
- KGK Science Inc., London, Ontario, Canada